CLINICAL TRIAL: NCT01620853
Title: Concordance Study for Detection of Chromosomal Aberrations Using FISH (ALK Test)in Non-small Cell Lung Cancer (NSCLC)
Brief Title: Detection of Chromosomal Aberrations in Non-small Cell Lung Cancer (NSCLC) Using Fluorescent in Situ Hybridization (FISH) (ALK Test)
Status: Completed | Type: Observational
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASI-ALK-F
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small cell lung cancer (NSCLC); ALK probe; FISH; Chromosomal aberrations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is the identification of chromosomal aberrations in non-small cell lung cancer (NSCLC) .

The imaging system is intended for diagnostic use as an aid to the pathologist in the detection, counting and classifying ALK FISH stained lung samples.

DETAILED DESCRIPTION:
The ALK Break Apart FISH test detects chromosomal aberrations via fluorescence in situ hybridization (FISH) in formalin-fixed paraffin-embedded (FFPE) non-small cell lung cancer (NSCLC) tissue specimens. The FDA approved ALK kit is designed to detect rearrangements involving the ALK gene (2p23). Results from the ALK Kit are intended for use, in conjunction with and not in lieu of current standard diagnostic procedures, as an aid for the pathologist in the identification of patients eligible for treatment with XALKORI® (crizotinib).

ELIGIBILITY:
Inclusion Criteria:

* Well stained slides with bright FISH signals

Exclusion Criteria:

* Very old slides that were already bleached

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having non-small cell lung cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
IVD study | 1 Day

CONTACTS AND LOCATIONS:
Locations (1):
- Scott & White Hospital,, Temple, Texas, United States